CLINICAL TRIAL: NCT05813418
Title: Identification of Predictive Biomarkers for Immune-Related Adverse Events (irAEs) in Patients
Brief Title: Identification of Predictive Biomarkers for Immune-Related Adverse Events (irAEs) in Patients Undergoing Immune CheckPoint Inhibitors (ICPI) Treatment
Acronym: Ibe2i-TIPCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Central Hospital Saint Quentin (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2019_843_0078
Record Dates: First submitted 2023-04-03; First posted 2023-04-14 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Immunotherapy; Immune Checkpoint Inhibitors; Immune-related Adverse Event; Predictive Biomarkers
Keywords: immunotherapy; immune checkpoint inhibitors; Immune-related Adverse Event; predictive biomarkers; plasmatic cytokines; circulating immune subpopulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: blood retriewal — blood retriewal for cytokine concentration measurement

SUMMARY:
In the last decades, cancer treatment was based on surgery, radiotherapy and chemotherapy.

Recently, treatments have largely evolved, first with targeted therapies (notably tyrosin kinase inhibitors, TKI) and then with immune checkpoint inhibitors (ICPI, notably anti-CTLA-4 and anti- PD1). The last ones can induce durable anti-tumoral responses in patients, even if metastases are present. Their mechanisms of action are focused on the activation of immune system in order to eliminate the tumor. ICPI, because of their mechanisms of action, target immune tolerance key components and can induce important immune toxicities (colitis, hepatitis, dermatitis, thyroiditis ...), leading to early discontinuation of treatment, severe or chronic morbidity, and can sometimes be lethal. It is of importance to detect patient at risk of irAEs, because of the increasing use of ICPI and the long- term response capacity in treated patients.

ELIGIBILITY:
Inclusion Criteria:

* patient with cancer, whatever initial tumoral histology and disease stage under ICPI treatment (anti-PD1 and/or anti-CTLA-4)
* age > 18
* followed in oncology, pneumology, dermatology, gastroenterology departments of Amiens-Picardie University Hospital or Saint Quentin hospital
* who received verbal and written information, and signed the consent form for the study

Exclusion Criteria:

* non ICPI treated patients
* patient who received a first line of ICPI treatment
* patient who received or is receiving MEK inhibitors as a treatment (because of possible lower response to ICPI treatment when associated)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-07-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Variation from baseline of IL6 concentration in riAEs patients | 6 months
  Variation from baseline of IL6 concentration (pG/mL) in riAEs patients
Variation from baseline of IL10 concentration in riAEs patients | 6 months
  Variation from baseline of IL10 concentration (pG/mL) in riAEs patients
Variation from baseline of IL15 concentration in riAEs patients | 6 months
  Variation from baseline of IL15 concentration (pG/mL) in riAEs patients
Variation from baseline of IL8 concentration in riAEs patients | 6 months
  Variation from baseline of IL8 concentration (pG/mL) in riAEs patients
Variation from baseline of INFgamma concentration in riAEs patients | 6 months
  Variation from baseline of INFgamma concentration (pG/mL) in riAEs patients
Variation from baseline of MCP-1 concentration in riAEs patients | 6 months
  Variation from baseline of MCP-1 concentration (pG/mL) in riAEs patients
Variation from baseline of MIP 1 alpha concentration in riAEs patients | 6 months
  Variation from baseline of MIP 1 alpha concentration (pG/mL) in riAEs patients
Variation from baseline of MIP 1 beta concentration in riAEs patients | 6 months
  Variation from baseline of MIP 1 beta concentration (pG/mL) in riAEs patients
Variation from baseline of sIL2R concentration in riAEs patients | 6 months
  Variation from baseline of sIL2R concentration (U/mL) in riAEs patients
Variation from baseline of sIL6R concentration in riAEs patients | 6 months
  Variation from baseline of sIL6R concentration (µG/mL) in riAEs patients

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No